CLINICAL TRIAL: NCT04295564
Title: Extending CPAP Therapy in Stable Preterm Infants to Increase Lung Growth and Function: A Randomized Controlled Trial
Brief Title: Extending CPAP Therapy in Stable Preterm Infants to Increase Lung Growth and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynthia McEvoy (Other)
Collaborators: Indiana University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Cynthia McEvoy, Principal Investigator, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eCPAP; R33HL147906 (NIH)
Record Dates: First submitted 2019-12-31; First posted 2020-03-04 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Neonatal; Premature Birth; Respiratory Distress Syndrome
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCPAP (Experimental): Participants will remain on CPAP for 2 additional weeks once CPAP stability criteria is met.
  Interventions: Other: Additional 2 weeks of CPAP
- dCPAP (No Intervention): Participants will discontinue CPAP as per usual care once CPAP stability criteria is met.

INTERVENTIONS:
Other: Additional 2 weeks of CPAP — Subjects will be randomized to an additional 2 weeks of CPAP vs. discontinuing CPAP per usual care.
  Arms: eCPAP

SUMMARY:
This is a study to see if an extra 2 weeks of continuous positive airway pressure (CPAP) in stable preterm infants in the neonatal intensive care unit (NICU) can cause increased lung growth and lung function in the infants as measured at 6 months of age by pulmonary function testing.

DETAILED DESCRIPTION:
This is a study to see if an extra 2 weeks of continuous positive airway pressure (CPAP) in stable preterm infants in the neonatal intensive care unit (NICU) can cause increased lung growth and lung function in the infants as measured at 6 months of age by pulmonary function testing. CPAP is a treatment widely used in the NICU in preterm infants right after they are born to help keep their lungs open/inflated. Although the benefit of CPAP after birth has been well studied, no one knows how long a stable preterm infant should stay on CPAP. The primary outcome of this study is to compare the lung volumes in the infants at 6 months of age by pulmonary function testing who were randomized to 2 extra weeks of CPAP in the NICU versus CPAP discontinuation, usual care. During the same pulmonary function test the investigators will also measure and compare how the infant's lungs diffuse gas.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at >24 to ≤ 32 weeks gestation
2. Treated with CPAP for ≥ 24 hours for respiratory distress (either as initial therapy or following extubation)

Exclusion Criteria:

1. Significant congenital heart disease
2. Major malformations
3. Chromosomal anomalies
4. Culture proven sepsis at consent
5. Complex maternal medical conditions
6. Clinical instability
7. Multiple gestations > twins
8. <3rd or >97th percentile for weight85
9. Participating in another neonatal randomized clinical trial with a competing outcome
10. Mother/legal guardian without stable method of communication

Ages: 1 Day to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy McEvoy, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Doernbecher Neonatal Care Center at Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual patient data related to primary outcome
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One year after publication of primary paper, lasting for 5 years.
Access Criteria: Signed data access agreement

REFERENCES:
- [Background] Lam R, Schilling D, Scottoline B, Platteau A, Niederhausen M, Lund KC, Schelonka RL, MacDonald KD, McEvoy CT. The Effect of Extended Continuous Positive Airway Pressure on Changes in Lung Volumes in Stable Premature Infants: A Randomized Controlled Trial. J Pediatr. 2020 Feb;217:66-72.e1. doi: 10.1016/j.jpeds.2019.07.074. Epub 2019 Sep 10. PMID 31519441
- [Background] Praca ELL, Tiller CJ, Kisling JA, Tepper RS. An alternative method to measure the diffusing capacity of the lung for carbon monoxide in infants. Pediatr Pulmonol. 2018 Mar;53(3):332-336. doi: 10.1002/ppul.23926. Epub 2017 Dec 19. PMID 29265767
- [Result] McEvoy CT, MacDonald KD, Go MA, Milner K, Harris J, Schilling D, Olson M, Tiller C, Slaven JE, Bjerregaard J, Vu A, Martin A, Mamidi R, Schelonka RL, Morris CD, Tepper RS. Extended Continuous Positive Airway Pressure in Preterm Infants Increases Lung Growth at 6 Months: A Randomized Controlled Trial. Am J Respir Crit Care Med. 2025 Apr;211(4):610-618. doi: 10.1164/rccm.202411-2169OC. PMID 39977011

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended Continuous Positive Airway Pressure (eCPAP): Participants will remain on continuous positive airway pressure (CPAP) for 2 additional weeks once CPAP stability criteria is met.
  Additional 2 weeks of CPAP: Subjects will be randomized to an additional 2 weeks of CPAP vs. discontinuing CPAP per usual care.
- Discontinue Continuous Positive Airway Pressure (dCPAP): Participants will discontinue CPAP as per usual care once CPAP stability criteria is met.
Period: Overall Study
Arm/Group | Extended Continuous Positive Airway Pressure (eCPAP) | Discontinue Continuous Positive Airway Pressure (dCPAP)
Started | 54 | 46
Completed | 53 | 46
Not Completed | 1 | 0
Not completed — Withdrawn by PI after discharge due to diagnosis of a rare chromosomal mutation. | 1 | 0

BASELINE CHARACTERISTICS:
Population: The number of infants who were randomized to extended CPAP (eCPAP) or discontinue CPAP (dCPAP) if they were > 24 and ≤ 32 weeks of gestational age, had required CPAP for ≥ 24 hours for clinical care, and when they met predefined respiratory stability criteria. 54 stable preterm infants were randomized to eCPAP and 46 stable preterm infants were randomized to dCPAP.
Groups:
- eCPAP: Participants randomized to stay on CPAP for 2 additional weeks once CPAP stability criteria were met.
- dCPAP: Participants randomized to discontinue CPAP once CPAP stability criteria were met.
- Total: Total of all reporting groups
Arm/Group | eCPAP | dCPAP | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Continuous [Mean (Standard Deviation); unit: weeks of postmenstrual age] | 32.4 (0.9) | 32.4 (0.8) | 32.4 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 35 | 22 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 9 | 28
  Not Hispanic or Latino | 34 | 37 | 71
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 42 | 33 | 75
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 54 | 46 | 100

OUTCOME MEASURES:

1. Primary Outcome: Alveolar Volume
Description: Establish that 2 additional weeks of CPAP in the NICU for stable preterm infants changes alveolar volume at approximately 6 months of age compared to infants who have CPAP discontinued, usual care. Measurements of alveolar volume were obtained at the same time as measurements of lung diffusion using an induced respiratory pause technique at an elevated lung volume of 30 cmH2O. During the passive expiration following the 4 second induced respiratory pause for gas exchange, carbon monoxide (CO) and helium (He) concentrations are used to calculate alveolar volume and lung diffusion. Results were expressed as averages of 2-3 measurements within 10%, adjusting for hemoglobin.
Time Frame: 4 - 8 months of age
Population: Decrease in the number of participants analyzed versus those initially randomized due to: Seven infants in the eCPAP arm did not complete VA testing due to the following reasons: 1 diagnosed with ARID1B mutation diagnosed after discharge and discontinued from study by the principal investigator; 1 with seizure disorder so could not be sedated; 3 mothers (one with a set of twins) refused sedation for the outpatient test; 1 infant with a technically unacceptable test.
Measure: Mean (Standard Error); unit: mL
Arm/Group | eCPAP | dCPAP
Number analyzed (Participants) | 47 | 46
mL | 500.2 (24.9) | 418.1 (23.4)
Statistical Analysis 1: Comparison: eCPAP vs dCPAP; Test type: Superiority; p < 0.05, Mixed Models Analysis — This is a calculate p value; adjusted for the correlation between twin pairs and gestational age at birth (stratification variable), sex, and length at outpatient testing; Mean Difference (Final Values) = 82.1, 95% CI 2-sided [8.3 to 155.9]

2. Secondary Outcome: Lung Diffusion
Description: Establish that 2 extra weeks of CPAP in stable preterm infants increases lung diffusion at approximately 6 months of age versus infants who have CPAP discontinued, usual care. Measurements of lung diffusion were obtained at the same time as measurements of alveolar volume using an induced respiratory pause technique at an elevated lung volume of 30 cmH2O. During the passive expiration following the 4 second induced respiratory pause for gas exchange, carbon monoxide (CO) and helium (He) concentrations are used to calculate alveolar volume and lung diffusion. Results were expressed as averages of 2-3 measurements within 10%, adjusting for hemoglobin.
Time Frame: 4 - 8 months of age
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL/min/mmHg
Arm/Group | eCPAP | dCPAP
Number analyzed (Participants) | 47 | 46
mL/min/mmHg | 3.4 (0.2) | 2.8 (0.1)
Statistical Analysis 1: Comparison: eCPAP vs dCPAP; Test type: Superiority; p < 0.02, Mixed Models Analysis — This is a calculated p value; Adjusted for correlation between twin pairs and gestational age at birth (stratification variable), sex, and length at outpatient test; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.1 to 1.1]

3. Secondary Outcome: Forced Expiratory Flows at 50% of the Expired Volume (FEF50)
Description: Establish that 2 extra weeks of CPAP in stable preterm infants increases forced expiratory flows at approximately 6 months of age versus infants who have CPAP discontinued, usual care. Forced expiratory flows were measured using the raised volume rapid thoracic compression technique following specific American Thoracic Society and European Respiratory Society criteria for acceptance.
Time Frame: 4 - 8 months of age
Population: Decrease in the number of participants analyzed versus those initially randomized due to: Infants in the eCPAP arm did not complete VA testing due to the following reasons: 1 diagnosed with ARID1B mutation diagnosed after discharge and discontinued from study by the principal investigator; 1 with seizure disorder so could not be sedated; 3 mothers (one with a set of twins) refused sedation for the outpatient test; and remainder with technically unacceptable test.
Measure: Mean (Standard Error); unit: mL/sec
Arm/Group | eCPAP | dCPAP
Number analyzed (Participants) | 38 | 38
mL/sec | 500.6 (18.2) | 437.9 (17.9)
Statistical Analysis 1: Comparison: eCPAP vs dCPAP; Test type: Superiority; p < 0.05, Mixed Models Analysis — This is a calculated p value; P-value adjusted for correlation between twin pairs and gestational age at birth (stratification variable), sex, and length at outpatient testing; Mean Difference (Final Values) = 62.7, 95% CI 2-sided [4.5 to 121]

4. Other Pre Specified Outcome: Number of Participants With the Occurrence of Wheeze
Description: Evaluate whether 2 extra weeks of CPAP in stable preterm infants results in lower respiratory morbidity through 12 months of age compared to infants who had CPAP discontinued, usual care. A standardized respiratory questionnaire was administered monthly through 12 months of age to ascertain this information on wheeze which was defined a priori.
Time Frame: through 12 months of age (+/- 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | eCPAP | dCPAP
Number analyzed (Participants) | 53 | 46
Participants | 23 | 26
Statistical Analysis 1: Comparison: eCPAP vs dCPAP; Test type: Superiority; p > 0.05, Regression, Logistic — This is a calculated p value; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.27 to 1.31]
Statistical Analysis 2: Comparison: eCPAP vs dCPAP; Test type: Superiority; p > 0.05, Regression, Logistic; Adjusted for gestational age at birth (stratification variable); Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.27 to 1.31]

5. Other Pre Specified Outcome: Bayley III Gross Motor Scores
Description: Evaluate whether 2 extra weeks of CPAP in stable preterm infants results in improved neurodevelopmental outcomes (Bayley III Gross Motor Scores) through 12 months of age compared to infants who had CPAP discontinued, usual care. These exams were performed by a licensed psychologist in the neurodevelopmental clinic.
Time Frame: through 12 months of age (+/- 2 months)
Reporting Status: Not Posted, anticipated posting 2025-10

ADVERSE EVENTS:
Time Frame: From consent through 12 months of age.
Description: Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | eCPAP | dCPAP
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/54 | 1/46
Other Adverse Events (participants affected / at risk) | 37/54 | 29/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eCPAP (N=54) | dCPAP (N=46)
Vocal cord paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Vocal cord paralysis on left post patent ductus arteriosus ligation. Determined to not be related to study.
streptococcus group B sepsis (Infections and infestations) | 1 (1) | 0 (0) — Streptococcus group B sepsis (late onset sepsis, requiring intubation). Determined not related to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eCPAP (N=54) | dCPAP (N=46)
Retinopathy of prematurity (Eye disorders) | 9 (9) | 5 (5)
Neonatal respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 6 (11)
Apnea neonatal (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 13 (18)
Feeding disorder NOS (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Nasal mucosal erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hemangioma of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Anemia of prematurity (Eye disorders) | 14 (14) | 9 (9)

LIMITATIONS AND CAVEATS:
Single center randomized controlled trial which may limit generalizability. Testing required mild sedation. Testing equipment is not commercially available. The study did not include preterm infants with the most severe respiratory disease. The clinical outcome of wheeze was obtained by parental report rather than assessment by medical personnel, which may have affected the accuracy of the wheeze outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT04295564/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT04295564/SAP_001.pdf